CLINICAL TRIAL: NCT03877939
Title: Detection of Kisspeptins and miRNAs in Patients With Non-viable Pregnancy
Acronym: TESTKM
Status: Completed | Type: Observational
Sponsor: Vida Recoletas Sevilla (Other)
Collaborators: IVI Madrid (Other); Instituto Valenciano de Infertilidad, IVI VALENCIA (Other); IVI Barcelona (Other)
Responsible Party: Sponsor
Other Study IDs: 1801-SEV-009-MF
Record Dates: First submitted 2019-03-14; First posted 2019-03-18 (Actual); Last update posted 2026-01-13 (Actual); Status verified 2026-01

CONDITIONS: Non-Viable Pregnancy
Keywords: Ectopic pregnancy; non-viable pregnancy; miRNA; Kisspeptin; β-HCG; biomarkers
MeSH Terms: conditions — Pregnancy, Ectopic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Peripheral blood samples will be collected to analyze:
  * Progesterone
  * miRNA-324-3p
  * Kisspeptin 54
  * KIR
  * HLA-C
  * miR-424-5p and miR-15b
  * Oral glucose tolerance test (OGTT)
  Additionaly, in patients with biochemical pregnancy, uterine biopsy samples will be collected to analyze:
  - miR-424-5p and miR-15b
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (5):
- Non-pregnant patients: Patients with β-hCG test < 10 UI/L.
  Interventions: Diagnostic Test: Blood samples collection for analysis
- Patients with viable pregnancy: Patients with β-hCG test > 10 UI/L whose pregnancy is confirmed between gestational weeks 6 and 8.
  Interventions: Diagnostic Test: Blood samples collection for analysis
- Patients with biochemical pregnancy: Patients with β-hCG test > 10 UI/L and without sac observed.
  Interventions: Diagnostic Test: Blood samples collection for analysis
- Patients with ectopic pregnancy: Patients with β-hCG test > 10 UI/L whose sac is implantated outside the uterine cavity.
  Interventions: Diagnostic Test: Blood samples collection for analysis
- Patients with clinical miscarriage: Patients with β-hCG test > 10 UI/L whose sac is implanted inside the uterine cavity, but non-viable pregnancy is confirmed before gestational week 8.
  Interventions: Diagnostic Test: Blood samples collection for analysis

INTERVENTIONS:
Diagnostic Test: Blood samples collection for analysis — Blood samples:
  Blood samples will be collected for the determination of the levels of various biomarkers (Kisspeptins and miRNAs), which are molecules that regulate the expression of proteins and can serve as markers for predicting pregnancy viability. Additionally, after biochemical or week 10 of clinical pregnancy confirmation, blood samples will be collected for KIR and HLA-C typing, Oral glucose tolerance test (OGTT) and analysis of the levels of miRNAs related with insulin resistance, miR-424-5p and miR-15b.
  Uterine biopsy (only in patients with BP):
  Uterine biopsy samples will be collected also after biochemical pregnancy confirmation for the determination of the levels of miRNAs related with insulin resistance, miR-424-5p and miR-15b.
  Other Names: Uterine biopsy sample collection (only in biochemical pregnancy patients)

SUMMARY:
Ectopic pregnancy (EP) is a pathology that affects 3%-16% of pregnancies in humans, being the main cause of morbidity and maternal mortality in the first trimester of pregnancy worldwide. The relevance of this problem has led to a demand on the scientific community, to obtain specific and early biomarkers in the determination of EP. In this context, the investigator's group has previously confirmed that both kisspeptin 54 and miR-324-3p are specific, selective and precise biomarkers to identify those patients suffering an EP. However, the utility of a diagnostic test using both biomarkers and other related ones in a population with other types of non-viable pregnancies should still be analysed.

DETAILED DESCRIPTION:
This is a pilot study in which we intend to determine the moment in which biomarkers begin to be detected in non-viable pregnancies, in order to subsequently be able to develop specific studies focused on that moment. The following visits will be required:

SCREENING VISIT: To be performed before β-hCG test. After recruitment and signing informed consent, patients will be assigned with a three-letter code identifying the clinic and three numbers indicating the order in which the patient is recruited by each clinic.

β-hCG VISIT: To be performed the day of the β-hCG test (week 4):

- Peripheral blood samples will be collected for Progesterone (P4), Kisspeptin 54 and miR-324-3p analysis.

In case of negative result, patient will be out of the study. In case of positive result, β-hCG test > 10 UI/L, patient will continue with the following visits.

SUBSEQUENT BLOOD EXTRACTION VISITS: To be performed on Mondays and Thursdays or Tuesdays and Fridays of each week from β-hCG test until non-viable pregnancy is confirmed or between weeks 6 and 8 when viable pregnancy is confirmed (a maximum of 10 blood sample extractions):

* Peripheral blood samples will be collected Progesterone (P4), Kisspeptin 54 and miR-324-3p will be analysed in these samples. Blood collection will be performed each day in a different arm, allowing a period between extractions in each arm of one week.
* In addition, an optional transvaginal ultrasound scan will be performed before each blood sample if patient wishes.

In case of pregnancy of unknown location (PUL), protocol will continue until VP or NVP is confirmed.

If NVP is confirmed before clinical pregnancy visit, patient will undergo an end of study visit.

CLINICAL PREGNANCY VISIT: To be performed between weeks 5+2 and 5+6, the same day that one of the subsequent blood extractions:

- A transvaginal ultrasound scan will be performed before the blood sample extraction.

In case of non-viable pregnancy, patient will perform the end of study visit. In case of clinical pregnancy, patient will continue with the following visits.

ONGOING PREGNANCY VISIT: To be performed between weeks 6 and 8, the same day that one of the subsequent blood extractions:

- A transvaginal ultrasound scan will be performed before the blood sample extraction. VP will be confirmed with this ultrasound scan.

In case of non-viable pregnancy, patient will undergo the end of study visit. In case of viable pregnancy, patient will undergo the end of study visit in week 10 of pregnancy.

END OF STUDY VISIT: To be performed after an ultrasound scan when NVP is confirmed or in week 10 of pregnancy. The following samples will be collected:

In case of ectopic pregnancy:

- Peripheral blood samples for Progesterone (P4), Kisspeptin 54 and miR-324-3p analysis.

In case of clinical miscarriage:

- Peripheral blood samples for Progesterone (P4), Kisspeptin 54 and miR-324-3p analysis.

In case of Biochemical pregnancy:

* Peripheral blood samples for Progesterone (P4), Kisspeptin 54 and miR-324-3p analysis.
* Blood sample for KIR typing.
* Blood samples of patient and partner for HLA-C typing. If partner does not attend to this visit, his sample may be collected in the following 3 weeks.
* Blood samples for detection of miRNAs related with insulin resistance, miR-424-5p and miR-15b.
* Oral glucose tolerance test (OGTT), including blood sample analysis before 75 g of glucose consumption and after 1h and 2 h.
* Uterine biopsy in the month in which the biochemical pregnancy is confirmed or in the following month (in P + 5) for detection of miRNAs related with insulin resistance, miR-424-5p and miR-15b.

In case of viable pregnancy in week 10 of gestation:

* Peripheral blood samples for Progesterone (P4), Kisspeptin 54 and miR-324-3p analysis.
* Blood sample for KIR typing.
* Blood samples of patient and partner for HLA-C typing. If partner does not attend to this visit, his sample may be collected in the following 3 weeks.
* Blood samples for detection of miRNAs related with insulin resistance, miR-424-5p and miR-15b.
* Data of an oral glucose tolerance test (OGTT) that patients perform routinely in the first trimester of pregnancy will be required.

ELIGIBILITY:
Inclusion Criteria:

* Patients who will perform SET.
* Patients using own oocytes.

Exclusion Criteria:

* Complicated uterine cavity.

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Those patient that have made a pre-embryonic transfer in the IVI RMA Seville, IVI RMA Madrid, IVI RMA Valencia, and IVI RMA Barcelona clinics will constitute patient population.
Sampling Method: Probability Sample
Enrollment: 433 (Actual)
Dates: Start 2019-09-15 (Actual); Primary Completion 2024-12-30 (Actual); Study Completion 2025-03-20 (Actual)

PRIMARY OUTCOMES:
Level of Kisspeptin 54 | Mar 2019 - Oct 2021
  Level in peripheral blood of Kisspeptin 54
Level of miR-324-3p | Mar 2019 - Oct 2021
  Level in peripheral blood of miR-324-3p

SECONDARY OUTCOMES:
Level of progesterone | Mar 2019 - Oct 2021
  Level in peripheral blood of progesterone
Level of hormone β-hCG | Mar 2019 - Oct 2021
  Level in peripheral blood of hormone β-hCG
Level of miRNAs related with insulin resistance, miR-424-5p and miR-15b | Mar 2019 - Oct 2021
  Level in peripheral blood of miR-424-5p and miR-15b in patients with viable and biochemical pregnancy
Level of miRNAs related with insulin resistance, miR-424-5p and miR-15b | Mar 2019 - Oct 2021
  Level in endometrial sample of miR-424-5p and miR-15b in patients with biochemical pregnancy
KIR typing | Mar 2019 - Oct 2021
  Killer-cell immunoglobulin-like receptors typing in patients with viable and biochemical pregnancy
HLA-C typing | Mar 2019 - Oct 2021
  HLA (human leucocyte antigens)-C typing in patients with viable and biochemical pregnancy and their partners
Oral glucose tolerance test (OGTT) | Mar 2019 - Oct 2021
  Including blood sample analysis before 75 g of glucose consumption and after 1h and 2 h.

CONTACTS AND LOCATIONS:
Overall Officials: Manuel Fernández-Sánchez, PhD, MD, Principal Investigator — IVI RMA Seville
Locations (2):
- Spain (2):
  - IVI RMA Madrid, Madrid, Madrid
  - IVI RMA Seville, Seville, Seville

IPD SHARING:
Plan to Share IPD: Undecided